CLINICAL TRIAL: NCT06981182
Title: EQUITy in Black Adult Health (EQUITA) - a Randomised Feasibility Trial of a Co-produced and Faith-placed Intervention to Increase Uptake of Breast, Cervical, Bowel, and AAA Screening in the North East of England, Leeds and Scotland
Brief Title: EQUITA - A Feasibility Trial of a Faith-placed Intervention to Increase Screening Uptake in Black Adults
Acronym: EQUITA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sunderland (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Floor Christie-de Jong, Associate Professor in Public Health for Medicine, University of Sunderland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIHR 164073; 164073 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2025-04-17; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Bowel Cancer; Cervical Cancer; Abdominal Aortic Aneurysm
Keywords: Cancer screening; Breast Cancer; Bowel Cancer; Cervical Cancer; Abdominal Aortic Aneurysm; Faith-placed intervention; Black adults; Randomised Controlled Trial; Feasibility study; Faith-based
MeSH Terms: conditions — Breast Neoplasms; Intestinal Neoplasms; Uterine Cervical Neoplasms; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person Workshop (Experimental): Participants will attend a co-produced 2-hour workshop delivered at a church at either sites; North East of England, Leeds and Scotland.
  Interventions: Other: Faith-placed intervention to promote breast, cervical, bowel, and AAA screening uptake in Black communities.
- No workshop (No Intervention): The control group will have regular church sessions and will be wait listed. They will receive the intervention after data collection is complete.

INTERVENTIONS:
Other: Faith-placed intervention to promote breast, cervical, bowel, and AAA screening uptake in Black communities. — The intervention includes a two-hour workshop, delivered in person to the entire congregation, that aims to promote the uptake of breast, cervical, bowel, and AAA screening among Black communities in the North East of England, Leeds and Scotland. However, we will only include effectiveness data (i.e., surveys and screening uptake) from those who meet the study eligibility criteria. The intervention will be a peer-led, multidimensional community workshop. It will incorporate multiple components that tackle barriers to screening and that are present in the existing IMCAN and PROCAN-B interventions, if the PICE group believe these are helpful, such as health education about breast, cervical, bowel and AAA screening delivered by a healthcare provider with an opportunity to ask questions, personal testimonials through survivors' stories, as well as members of the community discussing experiences of screening, and utilising community and peer support and religious leaders.
  Arms: In-person Workshop

SUMMARY:
The goal of this randomised feasibility trial is to examine feasibility and acceptability of a co-produced and faith-placed intervention to increase uptake of breast, cervical, bowel, and abdominal aortic aneurysm (AAA) screening among Black communities in the North East of England, Leeds and Scotland, United Kingdom (UK).

Participants will be invited to attend a two-hour workshop at each of the three study sites and will be randomly assigned to either the intervention group or the control group.

This 24-month feasibility study will inform the development of a full-scale randomised-controlled trial co-produced for Black people that uses culturally appropriate messages that support screening for early diagnosis in this underserved group.

DETAILED DESCRIPTION:
Over 2.4 million Black, Black British, Black Caribbean or African people live in the UK Black community, where lower screening rates place them at a higher risk of death due to lack of early diagnosis and provision of effective early treatment. Population health screening is largely under-researched in Black communities in the UK. Few studies have been conducted focusing on Black people and national screening programmes.

The EQUITA study builds on the IMCAN (Improving Muslim Women's CANcer Screening Uptake), and PROCAN-B ((Early diagnosis of PROstate CANcer for Black men) studies by using the same community-centred and participatory approach to apply a whole-community, multi-screening strategy to encourage uptake of breast, bowel, cervical, and AAA screening among Black communities. The intervention will retain the core elements of the participatory approach, including the Community Recruitment Leads on the research team, Public Involvement and Community Engagement (PICE) group for co-production, trained peer-facilitators, and faith-based engagement. The structured workshop format, which has demonstrated feasibility and acceptability in previous studies, will be tailored in collaboration with Black communities to ensure cultural relevance.

The study consists of six objectives with aligned work packages:

1. Can the existing intervention be adapted in partnership with a PICE group to improve engagement with breast, cervical, bowel, and AAA screening programmes in the Black community?
2. Can a two-arm cluster-randomised feasibility trial of the peer-led intervention be delivered in three sites: Leeds, North East of England and Scotland?
3. What are the perspectives of participants, peer facilitators, and key stakeholders on intervention and trial methodology, acceptability, and intervention implementation?
4. What is the feasibility trial's performance on key parameters and predefined progression criteria?
5. Is it feasible to conduct an economic evaluation to assess the cost-effectiveness of the intervention?
6. What are effective data dissemination strategies, and can the next phase be prepared by designing a study protocol for a definitive trial and logic model for implementation?

This feasibility trial will involve delivering a 2-hour workshop to 300 Black people (females aged 25-74 and males 50-74) in churches in Scotland, North East of England, and Leeds, who are either not or partially up to date with the screening they are eligible for. Participants will be randomly allocated to either the intervention or control group at each site. A process evaluation, including focus groups and stakeholder interviews, will guide modifications to the trial and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Members of participating churches (North East of England, Leeds, Scotland)
* Self-identify as Black,
* Female aged 25-74,
* Male aged 50-74,
* Not up to date with all screening tests for which they are eligible, e.g., women who are up to date with one form of screening (e.g., breast) will be eligible for recruitment if they are not up to date with others (e.g., cervical or bowel).

Exclusion Criteria:

* Not a member of participating churches (North East of England, Leeds, Scotland).
* Individuals who do not self-identify as Black
* Do not self-identity as Black
* Females aged outside the range of 25-74
* Males aged outside the range of 50-74.
* Individuals who are up to date with all screening tests for which they are eligible.

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Narrative description of feasibility | Month 1 - 24
  Using a mixed-methods approach and summarised as a narrative synthesis according to the progression criteria described below (Measures 1 - 11). Key feasibility domains include: time required for study setup and delivery; recruitment and retention of churches and participants; training and retention of peer facilitators; intervention delivery and adherence; data completeness and quality; and acceptability of procedures. Data sources will include recruitment and training logs, screening and consent forms, follow-up tracking sheets, and participant feedback surveys. Challenges and facilitators encountered will be documented in field notes by the study team. Quantitative data will be summarised descriptively (counts, percentages), and qualitative data will be thematically analysed. Findings will be assessed against pre-specified progression criteria to inform the viability of a future definitive trial.
(1) Number of churches recruited into the study | Month 3 - 7
  The number of churches recruited will be recorded using a site recruitment log maintained by the study team. This log will record church name, date of agreement to participate, and contact details of church representatives. Descriptive statistics (e.g., counts and percentages) will be used to summarise the data.
(2) Number of churches that consent to randomisation will be documented | Month 3 - 7
  A log will document the number of churches that agree to be randomised, including consent status and allocation group.
(3) Number of participants recruited | Month 3 - 7
  Participant screening and enrolment at baseline will be tracked in a participant recruitment log that includes date of screening, eligibility status, consent obtained (yes/no), and enrolment status. Numbers will be summarised using counts and percentages to assess recruitment feasibility.
(4) Distribution of recruited participants across age groups and screening programmes | Month 7 - 13
  Baseline demographic data (age, gender, and NHS screening eligibility) collected via participant questionnaires will be used to determine the distribution of participants across the four targeted screening programmes (cervical, breast, bowel, and AAA).
(5) Proportion of participants retained at 3-month follow up | Month 10 - 15
  A follow-up tracking log will record all participants due for 3-month follow-up, the mode of follow-up contact (e.g., phone, email), and whether data collection was completed. Retention rates will be calculated as the proportion of enrolled participants who complete the follow-up assessment.
(6) Acceptability of the informed consent procedures to participants | Month 10 - 18
  Acceptability of the informed consent process will be explored through qualitative interviews and/or focus groups conducted as part of the process evaluation. These discussions will examine participants' experiences of the consent process, including clarity of information, understanding of what participation involves, and overall satisfaction with how consent was obtained
(7) Suitability of data collection tools | Month 10 - 21
  Suitability of the data collection tools will be assessed through a mixed-methods approach. Completion rates will be calculated using descriptive statistics to evaluate the feasibility of administering the tools. In addition, feedback on the acceptability and clarity of the data collection measures will be gathered through qualitative methods (e.g. focus groups or interviews) and analysed thematically as part of the process evaluation.
(8) Proportion of participants providing consent to provide access to NHS screening data | Month 13 - 19
  The number of participants who explicitly consented to NHS data access will be recorded in the consent form and extracted into the study's NHS data access log. Percentages will be calculated relative to total enrolment. This will also be explored qualitatively
(9) Feasibility of accessibility of NHS screening data | Month 13 - 19
  Data request forms sub mitted to NHS and matched datasets returned will be tracked in a secure data access log. The proportion of successful data matches will be calculated in relative to total for unsuccessful data request submitted to NHS.
(10) Number of participants who become peer facilitators and time taken to train them | Month 4 - 13
  A training participation log will record the number of enrolled participants who registered for and attended peer facilitator training sessions. The number retained as peer facilitators at 3-month follow-up will also be recorded. Counts and retention percentages will be calculated.
  Dates of training registration, initiation, and completion will be documented in the training log. Time intervals will be calculated to determine the proportion trained within the target timeframe of 2-3 months.
(11) Acceptability of the intervention to participants | Month 10 - 18
  Qualitative feedback on the intervention will be collected post-intervention through focus groups and interviews with both intervention and control participants. Feedback will be summarised thematically.

SECONDARY OUTCOMES:
Attitude | Baseline (prior to intervention), Within 2 week post-intervention, 3 months post-intervention, 6 months post-intervention
  Change in attitude of barriers perceived towards screening programmes. This outcome is self-reported by participant
Religious Health Fatalism Questionnaire (RHFQ) | Baseline (prior to intervention)
  A questionnaire will be given to participants to test how religious beliefs influence health beliefs and willingness to obtain screening and medical treatments.
  RHFQ includes 8 statements that are answered on 5-point Likert scale: 1=strongly disagree, 2=disagree, 3=undecided, 4=agree, 5=strongly agree Total scores range from 8 to 40. Higher scores indicate higher levels of religious fatalism, thus a lower willingness to attend screening due to religious beliefs.
Modesty | Baseline (prior to intervention)
  The modesty measure for EQUITA is designed to assess the influence of cultural and religious values related to bodily privacy on cancer screening behaviours. Using two previously validated scales, the Modesty Measure for Muslim Women (MMM-W) by Padela et al. (2019) and Andrews' (2011) Modesty Scale.
  The measure comprises six items, rated on a 5-point Likert scale from Strongly Disagree (1) to Strongly Agree (5). Higher scores indicate stronger modesty beliefs related to bodily privacy. Scores will be analysed to examine the relationship between modesty and screening intentions or behaviours.
Socio-demographic Descriptions | Baseline (prior to intervention)
  Participant characteristics, such as age, location, education level, ethnicity, professional occupation and marital status, will be recorded and used for descriptive statistics ad subgroup analysis.
Cancer knowledge questions adapted from Cancer Awareness Measures (CAM) by Cancer Research UK | Baseline (prior to intervention), Within 2 week post-intervention, 3 months post-intervention, 6 months post-intervention
  The measure knowledge of symptoms and risk factors of breast, cervical, and bowel cancer, awareness of the NHS screening programmes including age of invitation and frequency, a question including 22 barriers to screening ranging from emotional to practical barriers, attitudinal change to screening, self-reported screening uptake, intention, preparedness, and sociodemographic descriptors. The CAM captures participants' socioeconomic status by measuring level of education, living arrangements (owning outright, mortgage, renting from local authority/privately, squatting, other), and their postcode. The questionnaire will be administered online through Qualtrics (a telephone option will also be offered). Most items are multiple-choice or Likert-scale. Higher scores indicate greater cancer knowledge. Total scores and subdomain scores will be compared over time.
AAA Knowledge Screening | Baseline (prior to intervention), Within 2 week post-intervention, 3 months post-intervention, 6 months post-intervention
  Questions assessing knowledge and awareness will be adapted from Suckow et al 2016These survey items, previously trialled in the UK and informed by other studies, include multiple-choice questions with single-choice responses on AAA definition, risk factors, detection methods, and the screening process. Correct responses will be summed. Higher scores indicate greater knowledge. Items are based on validated UK questionnaires.
Self-reported screening uptake | Baseline (prior to intervention), Within 2 week post-intervention, 3 months post-intervention
  Change in the number of participants who obtained screening following the intervention. This outcome is self-reported by participants. This (Yes/No) outcome will be assessed at follow-up. Uptake will be compared to baseline to assess the intervention's impact.
Actual screening uptake | 6 months post- intervention
  Screening data from the National Health Services (NHS) will be analysed to examine the change in the number of participants who obtained screening following the intervention.
Quality of life measure | Baseline (prior to intervention)
  Intervention participants will be asked to fill EQ-5D-5L questionnaires, which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems and 5 = extreme problems. Scores can be reported by individual dimension or as an index value (range: -0.281 to 1.0, where 1 = full health). Higher index scores represent better health-related quality of life.
Multimorbidity measure | Baseline (prior to intervention)
  Measures multimorbidity based on a disease count approach, which consists of a list of 35 conditions to be asked which they have, as well as the option to include any other conditions. The total number of conditions reported will be counted. Higher scores indicate greater multimorbidity.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - University of Glasgow, Glasgow, Scotland
  - Leeds Beckett University, Leeds
  - University of Sunderland, Sunderland

IPD SHARING:
Plan to Share IPD: No
IPD will not be publicly available, but may be shared upon reasonable request subject to data use agreements and ethics approval

REFERENCES:
- See also: NIHR Funding Award — https://www.fundingawards.nihr.ac.uk/award/NIHR164073